CLINICAL TRIAL: NCT07074054
Title: Early Anatomical and Functional Changes With Aflibercept 8 mg in Neovascular Age-Related Macular Degeneration: A Prospective Case Series
Brief Title: Aflibercept 8 mg for nAMD: Early Anatomical and Functional Changes
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, MD, PhD, Federico II University
Other Study IDs: 05809857 Federico II
Record Dates: First submitted 2025-06-17; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Presence of Retinal Fluid; Changes in Macular Pigment Optical Density
Keywords: nAMD; OCT; MPOD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients with naive nAMD treated with aflibercept 8 mg
- Control group: Patients with naive nAMD treated with aflibercept 2 mg

SUMMARY:
Neovascular age-related macular degeneration (nAMD) is one of the main causes of irreversible vision loss in older people worldwide.

the central role of vascular endothelial growth factor (VEFG) in the pathogenesis of nAMD has been extensively demonstrated. Since its introduction, intravitreal injection of targeted anti-VEGF antibodies has become the first-line treatment. Aflibercept 8 mg is a new formulation whose efficacy and safety as a new nAMD treatment has been demonstrated in the PULSAR study, emphasising its potential role in reducing the treatment burden in relation to the intended dosing intervals.

The aim of this study is to investigate early anatomical and functional changes in naïve nAMD patients treated with 8 mg aflibercept compared to patients treated with 2 mg aflibercept using OCT and MPOD, as potential parameters for functional outcome. To our knowledge, this is the first study to investigate these changes and the efficacy of aflibercept 8 mg as a potential fast-drying anti-VEGF treatment.

ELIGIBILITY:
Inclusion Criteria:

* age over 50 years; diagnosis of naïve nAMD due to the presence of active type 1 macular neovascularization (MNV)

Exclusion Criteria:

* previous ocular surgery, history of vitreoretinal and/or retinal vascular diseases, uveitis, myopia over 6 dioptres, significant corneal and/or lens opacity, glaucoma, ocular MNV related to other causes than nAMD, geographic atrophy, subretinal fibrosis, previous treatments for MNV

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients, over 50 years, diagnosed with naive nAMD, complicated by type 1 MNV, treated with aflibercept 8 mg
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
MPOD and OCT after aflibercept 8 mg loading phase | 7 months
  The parameters analyzed by OCT and MPOD 4 months after the treatment are: OCT and MPOD.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples, Federico II, Napoli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rinaldi M, Cennamo G, Concilio M, Corvino G, Riccardo A, Nubi R, Costagliola C. Aflibercept 8 mg in Neovascular AMD-A Fast-Drying Anti-VEGF Drug: A Prospective Morpho-Functional Pilot Study. Ophthalmol Ther. 2025 Dec 12. doi: 10.1007/s40123-025-01296-8. Online ahead of print. PMID 41388185